CLINICAL TRIAL: NCT05522829
Title: A Randomized, Double-blind Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of SCTV01E-1 (Alpha/Beta/Delta/Omicron (BA.1/BA.4/BA.5) Variants S-Trimer COVID-19 Vaccine) in Population Aged 18 Years and Older
Brief Title: A Study to Evaluate the Immunogenicity and Safety of a Recombinant Protein COVID-19 Vaccine SCTV01E-1 in Population Aged Above 18 Years
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCTV01E-1-UAE-1
Record Dates: First submitted 2022-08-30; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: SARS-CoV-2; COVID-19; vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Group SCTV01E-1 (Experimental): 3 doses of SCTV01E-1
  Interventions: Biological: SCTV01E-1 on D0; Biological: SCTV01E-1 on D28; Biological: SCTV01E-1 on D150
- Cohort 1: Group SCTV01E (Active Comparator): 3 doses of SCTV01E
  Interventions: Biological: SCTV01E on D0; Biological: SCTV01E on D28; Biological: SCTV01E on D150
- Cohort 2: Group SCTV01E-1 (Experimental): 2 doses of SCTV01E-1
  Interventions: Biological: SCTV01E-1 on D0; Biological: SCTV01E-1 on D120
- Cohort 2: Group SCTV01E (Active Comparator): 2 doses of SCTV01E
  Interventions: Biological: SCTV01E on D0; Biological: SCTV01E on D120

INTERVENTIONS:
Biological: SCTV01E-1 on D0 — Day 0; intramuscular injection
  Arms: Cohort 1: Group SCTV01E-1; Cohort 2: Group SCTV01E-1
Biological: SCTV01E-1 on D28 — Day 28; intramuscular injection
  Arms: Cohort 1: Group SCTV01E-1
Biological: SCTV01E-1 on D150 — Day 150; intramuscular injection
  Arms: Cohort 1: Group SCTV01E-1
Biological: SCTV01E on D0 — Day 0; intramuscular injection
  Arms: Cohort 1: Group SCTV01E; Cohort 2: Group SCTV01E
Biological: SCTV01E on D28 — Day 28; intramuscular injection
  Arms: Cohort 1: Group SCTV01E
Biological: SCTV01E on D150 — Day 150; intramuscular injection
  Arms: Cohort 1: Group SCTV01E
Biological: SCTV01E-1 on D120 — Day 120; intramuscular injection
  Arms: Cohort 2: Group SCTV01E-1
Biological: SCTV01E on D120 — Day 120; intramuscular injection
  Arms: Cohort 2: Group SCTV01E

SUMMARY:
The study is a randomized, double-blind Phase II study. It will evaluate the immunogenicity and safety of SCTV01E-1. Approximately 400 participants aged 18 years and older will be enrolled in this study. 160 participants who have not been vaccinated with any COVID-19 vaccine will be enrolled in Cohort 1 and randomly assigned to receive SCTV01E-1 or SCTV01E in a ratio of 1:1. 240 participants who were fully vaccinated with 2 or 3 doses of inactivated COVID-19 vaccines at least three months ago will be enrolled in Cohort 2 and randomly assigned to receive SCTV01E-1 or SCTV01E in a ratio of 1:1.

DETAILED DESCRIPTION:
The study is a randomized, double-blind Phase II study. It will evaluate the immunogenicity and safety of SCTV01E-1. Approximately 400 participants aged 18 years and older will be enrolled in this study.

160 participants who have not been vaccinated with any COVID-19 vaccine will be enrolled in Cohort 1 and randomly assigned to the Group SCTV01E-1 and Group SCTV01E in a ratio of 1:1. All participants will receive 3 doses of vaccinations: Vaccination 1 on D0, Vaccination 2 on D28 and Vaccination 3 on D150. Participants in Group SCTV01E-1 will receive 3 doses of SCTV01E-1, and participants in Group SCTV01E will receive 3 doses of SCTV01E.

240 participants who were fully vaccinated with 2 or 3 doses of inactivated COVID-19 vaccines at least three months ago will be enrolled in Cohort 2 and randomly assigned to Group SCTV01E-1 and Group SCTV01E in a ratio of 1:1. All participants will receive 2 doses of vaccinations: Vaccination 1 on D0 and Vaccination 2 on D120. Participants in Group SCTV01E-1 will receive 2 doses of SCTV01E-1, and participants in Group SCTV01E will receive 2 doses of SCTV01E.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years when signing ICF;
2. For Cohort 1: Participants who have not been vaccinated with any COVID-19 vaccine; For Cohort 2: Participants who were fully vaccinated with 2 or 3 doses of inactivated COVID-19 vaccine and the interval between the last dose of previously vaccination and the 1st study vaccination is 3 to 24 months;
3. Healthy participants or participants with pre-existing medical conditions that are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, chronic cholecystitis and cholelithiasis, chronic gastritis, etc. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization as a consequence of worsening disease state for at least 3 months prior to study participation;
4. The participant or his/her legal representative can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that are available if they do not participate in the trial;
5. The participant can read, understand, and fill in record cards by himself/herself or with help;
6. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the last dose of study vaccination.

Exclusion Criteria:

1. Presence of fever (oral temperature ≥37.5℃) within 3 days before the 1st study vaccination;
2. For Cohort 2 only: Known history of COVID-19 or asymptomatic SRAS-CoV-2 infection;
3. A history of allergic reactions to any vaccines or drugs, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
4. Immunocompromised patients suffering from immunodeficiency diseases, significant diseases, or immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc;
5. Long-term use of immunosuppressant therapy or immunomodulatory drugs for >14 days within the six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
6. Those who have a history of HIV or tested positive for HIV;
7. For Cohort 1, participants received any drugs or vaccines used to prevent COVID-19; for Cohort 2, participants received other drugs or vaccines used to prevent COVID-19 besides inactivated COVID-19 vaccines;
8. A history of Severe Acute Respiratory Syndrome (SARS), Middle East Respiratory Syndrome (MERS), or related vaccination;
9. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
10. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (skin basal cell carcinoma and carcinoma in-situ of cervix are exceptions and will not be excluded), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
11. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
12. Patients on antituberculosis therapy;
13. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
14. Participants who received other investigational drugs within 1 month before the study vaccination;
15. Participants who have acute illness, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
16. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
17. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
18. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
19. Those who plan to donate ovum or sperms during the study period;
20. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
21. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse or confound the study results, or non-conformance with the maximal benefits of the participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Geometric mean titers (GMT) of neutralizing antibodies (nAb) against Omicron subvariant (BA.5) on Day 42. | Day 42 after the study vaccination
Cohort 1: Geometric mean titers (GMT) of neutralizing antibodies (nAb) against Omicron subvariant (BA.5) on Day 178. | Day 178 after the study vaccination
Cohort 2: Geometric mean titers (GMT) of neutralizing antibodies (nAb) against Omicron subvariant (BA.5) on Day 28. | Day 28 after the study vaccination
Cohort 2: Geometric mean titers (GMT) of neutralizing antibodies (nAb) against Omicron subvariant (BA.5) on Day 148. | Day 148 after the study vaccination

SECONDARY OUTCOMES:
Cohort 1: Seroresponse rates of nAb against Omicron subvariant (BA.5) on Day 42. | Day 42 after the study vaccination
Cohort 1: Seroresponse rates of nAb against Omicron subvariant (BA.5) on Day 178. | Day 178 after the study vaccination
Cohort 1: Incidence and severity of solicited AEs within 7 days after each of the study vaccination. | Day 0 to Day 7 after each of the study vaccination
Cohort 1: Incidence and severity of unsolicited AEs within 28 days after each of the study vaccination. | Day 0 to Day 28 after each of the study vaccination
Cohort 1: Incidence and severity of SAEs and AESIs within 180 days after each of the study vaccination. | During the whole study
Cohort 2: Seroresponse rates of nAb against Omicron subvariant (BA.5) on Day 28. | Day 28 after the study vaccination
Cohort 2: Seroresponse rates of nAb against Omicron subvariant (BA.5) on Day 148. | Day 148 after the study vaccination
Cohort 2: Incidence and severity of solicited AEs within 7 days after each of the study vaccination. | Day 0 to Day 7 after each of the study vaccination
Cohort 2: Incidence and severity of unsolicited AEs within 28 days after each of the study vaccination. | Day 0 to Day 28 after each of the study vaccination
Cohort 2: Incidence and severity of SAEs and AESIs within 180 days after each of the study vaccination. | During the whole study